CLINICAL TRIAL: NCT02600026
Title: Video Feedback Intervention for Cognitively Impaired Older Drivers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Brian Ott, Brian R. Ott, MD, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 799824-2
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Impaired Driving

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video Camera: Intervention (Experimental): DriveCam video event recorder with feedback
  Interventions: Device: DriveCam; Behavioral: Feedback
- Video Camera: Monitoring (Placebo Comparator): DriveCam video event recorder with no feedback
  Interventions: Device: DriveCam

INTERVENTIONS:
Device: DriveCam — Video event monitoring device
Behavioral: Feedback — Video feedback intervention
  Arms: Video Camera: Intervention

SUMMARY:
This study will use an in-car monitoring system supplemented with video feedback to reduce the number of unsafe driving behaviors. If successful, this technology will provide a means to enhance public safety on the roads that could be adopted immediately in this at-risk group of drivers. The intervention will also maximize the time for independent driving, improving the overall quality of life of these individuals.

DETAILED DESCRIPTION:
The goals of this clinical trial are to 1) document real-time impaired driving behaviors, and 2) reduce their occurrence, to improve the safety of cognitively impaired elders who continue to drive. This will be accomplished by placing small digital video event recording devices in the vehicles of 60 older cognitively impaired drivers. A 3-month baseline will establish the frequency of unsafe driving events, followed by a 3-month video feedback intervention during which the driver and family member will review the video recorded errors on a weekly basis. Active treatment will be compared to video monitoring with no feedback. A 6-month post-intervention phase will establish sustainability of the treatment.

The results of this clinical trial will confirm the potential to improve driving safety among older drivers with cognitive impairment using a behavior modification approach aimed directly at the problem behaviors observed in their natural driving environment. Knowledge gained about the magnitude and duration of the treatment effect and the potential of using an internet based feedback program will provide the impetus to optimize and ultimately implement the intervention to improve the safety of older drivers with mild cognitive impairment and early AD.

ELIGIBILITY:
Inclusion Criteria:

* age 50-90
* will be categorized as CDR= 0.5, or 1
* English speaking
* currently driving adults
* have a valid driving license
* have at least 10 years of driving experience
* have a MMSE < 28
* have an adult family member or other caregiver, age >21, to participate in video feedback

Exclusion Criteria:

* ophthalmologic, physical, or neurologic disorders other than dementia that impair their driving abilities
* visual acuity worse than 20/40 in best eye using distance vision measured by wall chart
* homonymous hemianopia or bitemporal hemianopia
* musculoskeletal disorders causing major physical handicaps
* history of alcohol or substance abuse by DSM V criteria within the past year
* sedating medications that impair level of consciousness or attention
* language impairment that would interfere with the ability to participate in the educational intervention
* previous road test evaluation or opinion of caregiver or health professional that participant is unsafe to drive.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of unsafe driving events | 9 months
  Unsafe events rated as > 5 points using a modification of standard scale developed by Drivecam monitoring video service. This includes incidents, near-crashes, and crashes, sub classified as being triggered by hard turns, severe braking, and/or impact, adjusted for miles driven.

SECONDARY OUTCOMES:
Severity score of unsafe driving events | 9 months
  Measured by sum of all demerit points for events rated >5 adjusted for miles driven, during intervention and 6-month follow-up. The severity rating score derived and reported by DriveCam experts has been previously used in a longitudinal study of ambulance drivers demonstrating reduction in not only events, but also severity scores for events, as well as our own feasibility study. This measure will provide additional evidence supporting improvement in safe driving for our intervention trial. To demonstrate safe driving as an outcome, one would like to show not only a reduction in frequency of events, but also a reduction in the severity of those driving errors.
Time to driving cessation | 1-2 years
  Time to driving cessation (e.g., due to road-test failure, at-fault motor vehicle accident, cognitive decline progression) measured over one to two years from baseline. Information on time to driving cessation, i.e., "driving retirement," will be obtained from annual telephone follow-up calls to the driving participant and family member up to the end of the 3-year study period.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ott, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States